CLINICAL TRIAL: NCT02547844
Title: Open Randomized Study to Assess the Evolution of Plasma Lipid Profile by Lipidomic in Patients Infected With Human Immunodeficiency Virus (HIV-1) With Viral Suppression That Change Atripla® to Eviplera® Compared to Continue With Atripla®
Brief Title: Evolution of Plasma Lipid Profile in Patients With HIV1 Who Change Atripla to Eviplera Compared to Continue With Atripla
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EfaRiLipidomics
Record Dates: First submitted 2015-09-10; First posted 2015-09-11 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: HIV-1
MeSH Terms: interventions — efavirenz; Emtricitabine; Tenofovir; Efavirenz, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Rilpivirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- efavirenz + emtricitabina + tenofovir (Active Comparator): Patients assigned to the control group will continue receiving the same medication than before to be included in the study: Atripla (efavirenz + emtricitabina + tenofovir)
  Interventions: Drug: efavirenz + emtricitabina + tenofovir
- rilpivirina + emtricitabina + tenofovir (Experimental): Patients assigned to the experimental group will change the medication that are taking before to enter in the study ( atripla) for eviplera (rilpivirina + emtricitabina + tenofovir)
  Interventions: Drug: rilpivirina + emtricitabina + tenofovir

INTERVENTIONS:
Drug: efavirenz + emtricitabina + tenofovir
  Other Names: atripla
  Arms: efavirenz + emtricitabina + tenofovir
Drug: rilpivirina + emtricitabina + tenofovir
  Other Names: eviplera
  Arms: rilpivirina + emtricitabina + tenofovir

SUMMARY:
To compare the lipidomic profile in patients with HIV-1 with viral suppression changing efavirenz + emtricitabine + tenofovir (Atripla) to rilpivirine + emtricitabine + tenofovir (Eviplera®) versus a group of patients that continue with Atripla®.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or above
* Patients infected with HIV-1
* Patients treated with Atripla at least the last 6 months.
* Patients with virologic suppression (HIV RNA <50 copies / ml) for at least the last 6 months.
* Women of childbearing potential must use contraception double barrier.
* Voluntary signature of informed consent

Exclusion Criteria:

* Any acute or chronic (besides chronic HIV-1) disease that could interfere with the analysis of lipidomic
* Women pregnant or lactating
* Abuse of alcohol or other drugs
* Body Mass Index (BMI)> 25
* Use of drugs that may affect lipid metabolism (lipid-lowering drugs, steroids ...)
* Patients unable to understand the study protocol or any other condition that in the investigator's opinion could jeopardize compliance with the protocol
* History or presence of allergy to any of the study drugs or their components

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-09; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Changes in plasma lipid profile measured by lipidomic in patients with chronic HIV-1 with antiretroviral therapy and viral suppression. | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Vall d'Hebron, Barcelona, Spain